CLINICAL TRIAL: NCT02956850
Title: A Phase I, Sponsor-Open, Investigator-Blinded, Subject-Blinded, Multi-Center, Placebo-Controlled Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral Administration of RO7020531: (1). Single and Multiple Ascending Doses in Healthy Male and Female Subjects; (2). 6-week Treatment of Patients With Chronic Hepatitis B Virus Infection
Brief Title: A Study in Healthy Volunteers and in Participants With Chronic Hepatitis B to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of RO7020531
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP39305; 2016-003723-38 (EudraCT Number)
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — RO7020531

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Part I: SAD in Healthy Volunteers (Experimental): Healthy volunteers will receive single dose of RO7020531 or matching placebo orally on Day 1 of each cohort. A planned dose-escalation sequence for SAD is 3 milligrams (mg), 10 mg, 20 mg, 40 mg, 60 mg, 100 mg, 140 mg, and 170 mg.
  Interventions: Other: Placebo; Drug: RO7020531
- Part I: MAD in Healthy Volunteers (Experimental): Healthy volunteers will receive RO7020531 (100 mg, 140 mg, and 170 mg as selected based on safety, pharmacokinetic (PK) and pharmacodynamic (PD) data of SAD cohorts) or matching placebo orally every other day (QOD) from Day 1 through to Day 13.
  Interventions: Other: Placebo; Drug: RO7020531
- Part II: CHB Participants (Experimental): CHB participants will receive RO7020531 (150 mg and 170 mg as selected based on safety, PK and PD data of MAD cohorts) or matching placebo orally QOD from Day 1 through to Day 41, unless in Cohort 4 in case of once a week (QW) dosing as dose modification.
  Interventions: Other: Placebo; Drug: RO7020531

INTERVENTIONS:
Other: Placebo — Placebo matching to RO7020531 will be administered as per schedule specified in the respective arm.
Drug: RO7020531 — RO7020531 will be administered as per schedule specified in the respective arm.

SUMMARY:
This sponsor-open, investigator- and participant-blinded, multi-center study will assess the safety, tolerability, pharmacokinetics and pharmacodynamics of RO7020531 in healthy participants and in participants with chronic hepatitis B. Part I will be conducted in two portions: Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) which will include only healthy volunteers. Part II will commence after completion of the MAD portion of Part I and will include only Chronic Hepatitis B (CHB) participants.

ELIGIBILITY:
Inclusion Criteria:

Part 1: SAD and MAD in Healthy Volunteers

* Non-smokers, or use of less than (<) 10 cigarettes (or equivalent nicotine-containing product) per day
* Negative Anti-Nuclear Antibody (ANA) test; or positive with dilutions not greater than 1:40 and with no associated history or symptoms of potential connective tissue disease or other immune-mediated diseases

Part 2: CHB Participants

* CHB infection (positive test for Hepatitis B surface antigen [HBsAg] for more than 6 months prior to randomization)
* For Cohort 1, 2, 3 and 4: HBsAg detectable at screening
* For Cohort 1, 2 and 3: Hepatitis B virus deoxyribose nuclic acid (HBV DNA) < 90 international unit per milliliter (IU/mL) for at least 6 months prior to randomization; HBV DNA < 90 IU/mL at screening by Roche Cobas assay
* For Cohort 4: HBV DNA at screening >= 2 × 10*4 IU/mL for HBeAg positive and >= 2 x 10*3 IU/mL for hepatitis B e antigen (HBeAg) negative participants
* For Cohort 1, 2 and 3: Alanine amino transferase (ALT) =<1.5 × upper limit of normal (ULN) during the 6 months prior to randomization confirmed by two measurements separated by at least 14 days; ALT at screening =< 1.5 × ULN.
* For Cohort 4: ALT and aspartate aminotransferase (AST) at screening and Day -1 visit: =< 5 × ULN.
* Negative ANA test; or positive with dilutions not greater than 1:40 and with no associated history or symptoms of potential connective tissue disease or other immune-mediated diseases
* Liver biopsy, Fibroscan® or equivalent elastography test obtained within 6 months prior to randomization demonstrating liver disease consistent with chronic HBV infection with absence of cirrhosis and absence of extensive bridging fibrosis (cirrhosis or extensive bridging fibrosis are defined as greater than or equal to (>/=) Metavir 3, recommended cut-off for Fibroscan 8.5 kilopascals [kPa])
* For Cohort 1, 2 and 3: On treatment with tenofovir, entecavir, adefovir, or telbivudine, either as single agents or in combination, for at least 6 months
* For Cohort 4: Hepatitis B virus (HBV) treatment naïve or not on any anti-HBV treatment for the past 6 months

Exclusion Criteria:

Part 1: SAD and MAD in Healthy Volunteers

* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune haemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis, multiple sclerosis, or any other autoimmune disease); clinically significant psychiatric disease, acute infection (e.g., influenza), gastrointestinal (GI) disease (including inflammatory bowel disease, peptic ulcer disease, GI hemorrhage)
* History of having received or currently receiving any systemic anti-neoplastic (including radiation) or immune-modulatory treatment (including systemic oral or inhaled corticosteroids, IFN or pegylated interferon [PEG-IFN]) within the 8 weeks prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
* Any clinically significant concomitant disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study
* Positive Hepatitis A virus antibody (HAV Ab IgM), HBsAg, Hepatitis C antibody (HCV Ab), or positive for human immunodeficiency virus (HIV) at screening
* History of clinically significant thyroid disease; also, participants with clinically significant elevated thyroid-stimulating hormone (TSH) concentrations at screening
* Positive results for anti-mitochondrial antibody (AMA), anti-smooth muscle antibody (ASMA) or thyroid peroxidase antibody

Part 2: CHB Participants

* History of liver cirrhosis
* History or other evidence of bleeding from esophageal varices
* Decompensated liver disease (e.g., Child-Pugh Class B or C clinical classification or clinical evidence such as ascites or varices)
* History or other evidence of a medical condition associated with chronic liver disease other than HBV infection (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposure, thalassemia, nonalcoholic steato-hepatitis, etc.). A clinical diagnosis of fatty liver is allowed provided that non alcoholic steatohepatitis (NASH) has been excluded by liver biopsy.
* Documented history or other evidence of metabolic liver disease within one year of randomization
* Positive test for Hepatitis A virus (IgM anti-HAV), Hepatitis C virus (HCV), Hepatitis D virus, Hepatitis E virus (HEV), or human immunodeficiency virus (HIV).
* History of or suspicion of hepatocellular carcinoma or alpha fetoprotein >/=13 nanograms per milliliter (ng/mL) at screening
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune haemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis, multiple sclerosis, or any other autoimmune disease); clinically significant psychiatric disease; acute infection (e.g., influenza); GI disease (including inflammatory bowel disease, peptic ulcer disease, GI hemorrhage, or history of pancreatitis); clinically significant cardiovascular (including postural hypotension), endocrine, renal, ocular, pulmonary or neurological disease.
* History of having received or currently receiving any systemic anti-neoplastic (including radiation) or immune-modulatory treatment (including systemic oral or inhaled corticosteroids,IFN or PEG-IFN) within the 8 weeks prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
* Cohort 4: Concurrent HBV treatments
* History of organ transplantation
* Clinically significant thyroid disease; also, participants with clinically significant elevated TSH concentrations at screening
* Positive results for AMA, ASMA or thyroid peroxidase antibody

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Bulgaria (2):
  - Gastroenterology department, Second clinic of internal diseases, Sofia
  - COMAC Medical; Clinical Research Unit for Phase I, Sofia
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - The Chinese University of Hong Kong, Shatin
- Italy (3):
  - Azienda Ospedaliero Universitaria Di Modena Policlinico; U.O. Farmacia, Modena, Emilia-Romagna
  - ASST PAPA GIOVANNI XXIII; Epatologia e gastroenterologia pediatrica e dei trapianti, Bergamo, Lombardy
  - Medicina Generale ed Epatologia (Humanitas-Rozzano), Rozzano, Lombardy
- Academisch Medisch Centrum Universiteit Amsterdam; Dermatology and VU University Medical Center, Amsterdam, Netherlands
- Auckland Clinical Studies, Auckland, New Zealand
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
  - Taichung Veterans General Hospital, Xitun Dist.
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- United Kingdom (2):
  - Royal Liverpool University Hospital, Liverpool
  - King College Hospital NHS Foundation Trust, London

REFERENCES:
- [Derived] Yuen MF, Balabanska R, Cottreel E, Chen E, Duan D, Jiang Q, Patil A, Triyatni M, Upmanyu R, Zhu Y, Canducci F, Gane EJ. TLR7 agonist RO7020531 versus placebo in healthy volunteers and patients with chronic hepatitis B virus infection: a randomised, observer-blind, placebo-controlled, phase 1 trial. Lancet Infect Dis. 2023 Apr;23(4):496-507. doi: 10.1016/S1473-3099(22)00727-7. Epub 2022 Dec 9. PMID 36509100

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 16 investigative sites in New Zealand, Hong Kong, Thailand, Taiwan, New Zealand, Bulgaria, United Kingdom, Italy and Netherlands from 12 December 2016 to 15 June 2021.
Pre-assignment Details: A total of 160 participants were enrolled in the study. 110 participants were enrolled in Part 1 and 50 participants were enrolled in Part 2.
Groups:
- Part 1 Cohorts 1-8, Single Ascending Dose (SAD): Placebo: In SAD Cohorts 1-8, sixteen healthy volunteers (HVs), two in each cohort, received a single dose of RO7020531 matching placebo, on Day 1
- Part 1 SAD: Cohort 1: HVs received single dose of RO7020531, 3 milligrams (mg), orally on Day 1.
- Part 1 SAD: Cohort 2: HVs received single dose of RO7020531, 10 mg, orally on Day 1.
- Part 1 SAD: Cohort 3: HVs received single dose of RO7020531, 20 mg, orally on Day 1.
- Part 1 SAD: Cohort 4: HVs received single dose of RO7020531, 40 mg, orally on Day 1.
- Part 1 SAD: Cohort 5: HVs received single dose of RO7020531, 60 mg, orally on Day 1.
- Part 1 SAD: Cohort 6: HVs received single dose of RO7020531, 100 mg, orally on Day 1.
- Part 1 SAD: Cohort 7: HVs received single dose of RO7020531, 140 mg, orally on Day 1.
- Part 1 SAD: Cohort 8: HVs received single dose of RO7020531, 170 mg, orally on Day 1.
- Part 1 Cohorts 1-3, Multiple Ascending Dose (MAD): Placebo: In MAD Cohorts 1,2, and 3, six HVs, two in each cohort, received RO7020531 matching placebo orally on Day 1 and every other day (QOD) for 13 days.
- Part 1 MAD: Cohort 1: HVs received RO7020531, 100 mg, orally, on Day 1 and QOD for 13 days.
- Part 1 MAD: Cohort 2: HVs received RO7020531, 140 mg, orally, on Day 1 and QOD for 13 days.
- Part 1 MAD: Cohort 3: HVs received RO7020531, 170 mg, orally, on Day 1 and QOD for 13 days.
- Part 2 Cohorts 1-3: Placebo: In Cohorts 1,2, and 3, six participants, two in each cohort, Participants received RO7020531 matching placebo, along with nucleoside/nucleotide analogue (NUC) treatment, orally, on Day 1 and QOD for 41 days.
- Part 2: Cohort 1 and 2: Sixteen participants received RO7020531, 150 mg, along with NUC treatment, orally, on Day 1 and QOD for 41 days. Cohorts 1 and 2 were both 150 mg cohorts and was presented as a single dose group.
- Part 2: Cohort 3: Participants received RO7020531, 170 mg, along with NUC treatment, orally, on Day 1 and QOD for 41 days.
- Part 2 Cohort 4: Placebo: Treatment naive participants received RO7020531 matching placebo, orally, on Day 1 and QOD for 41 days.
- Part 2: Cohort 4: Treatment naive participants received RO7020531, 150 mg, orally, on Day 1 and QOD for 41 days.
Period: Overall Study
Arm/Group | Part 1 Cohorts 1-8, Single Ascending Dose (SAD): Placebo | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8 | Part 1 Cohorts 1-3, Multiple Ascending Dose (MAD): Placebo | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3 | Part 2 Cohorts 1-3: Placebo | Part 2: Cohort 1 and 2 | Part 2: Cohort 3 | Part 2 Cohort 4: Placebo | Part 2: Cohort 4
Started | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 8 | 8 | 6 | 16 | 8 | 5 | 15
Completed | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 8 | 8 | 6 | 16 | 8 | 5 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who had received at least 1 dose of the study drug.
Groups:
- Part 1 Cohorts 1-8 SAD: Placebo: In SAD Cohorts 1-8, sixteen HVs, two in each cohort, received a single dose of RO7020531 matching placebo, on Day 1.
- Part 1 SAD: Cohort 1: HVs received single dose of RO7020531, 3 mg, orally on Day 1.
- Part 1 Cohorts 1-3, MAD: Placebo: In MAD Cohorts 1,2, and 3, six HVs, two in each cohort, received RO7020531 matching placebo orally on Day 1 and QOD for 13 days.
- Part 2 Cohorts 1-3: Placebo: In Cohorts 1,2, and 3, six participants, two in each cohort, Participants received RO7020531 matching placebo, along with NUC treatment, orally, on Day 1 and QOD for 41 days.
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohorts 1-8 SAD: Placebo | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8 | Part 1 Cohorts 1-3, MAD: Placebo | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3 | Part 2 Cohorts 1-3: Placebo | Part 2: Cohort 1 and 2 | Part 2: Cohort 3 | Part 2 Cohort 4: Placebo | Part 2: Cohort 4 | Total
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 8 | 8 | 6 | 16 | 8 | 5 | 15 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (10.1) | 31.5 (15.8) | 37.6 (16.2) | 22.6 (2.7) | 23.8 (4.5) | 29.3 (7.0) | 33.4 (12.5) | 25.8 (3.5) | 29.5 (10.9) | 27.2 (4.0) | 26.8 (3.9) | 26.5 (2.9) | 25.0 (7.5) | 49.3 (13.3) | 47.6 (8.9) | 42.4 (10.5) | 42.6 (11.5) | 40.1 (9.3) | 33.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 2 | 2 | 2 | 1 | 3 | 2 | 2 | 2 | 4 | 2 | 1 | 4 | 2 | 1 | 9 | 48
  Male | 11 | 6 | 6 | 6 | 6 | 6 | 7 | 5 | 6 | 4 | 6 | 4 | 6 | 5 | 12 | 6 | 4 | 6 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Not Hispanic or Latino | 14 | 8 | 7 | 8 | 8 | 7 | 7 | 7 | 8 | 6 | 8 | 8 | 8 | 6 | 15 | 8 | 5 | 14 | 152
  Not Stated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 2 | 1 | 0 | 2 | 1 | 3 | 1 | 4 | 0 | 0 | 3 | 2 | 1 | 9 | 5 | 2 | 6 | 44
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
  Native Hawaiian or other Pacific Islander | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 7
  White | 13 | 4 | 6 | 8 | 6 | 7 | 5 | 7 | 3 | 6 | 7 | 4 | 4 | 4 | 5 | 3 | 3 | 8 | 103
  Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of SAD Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation healthy volunteer (HV)/participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product, any new disease or exacerbation of an existing disease (a worsening in the character, frequency, or severity of a known condition and recurrence of an intermittent medical condition (e.g., headache) not present at baseline.
Time Frame: From randomization up to Day 29
Population: Safety analysis population included all HVs who had received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-8 SAD: Placebo | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
percentage of participants | 31.3 | 25.0 | 50.0 | 25.0 | 25.0 | 25.0 | 25.0 | 25.0 | 37.5

2. Primary Outcome: Part 1: Percentage of MAD Participants With AEs
Description: as for outcome 1
Time Frame: From randomization up to Day 41
Population: Safety analysis population included all HVs who had received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-3, MAD: Placebo | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 6 | 8 | 8 | 8
percentage of participants | 83.3 | 75.0 | 87.5 | 87.5

3. Primary Outcome: Part 2: Percentage of Chronic Hepatitis B Participants With AEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product, any new disease or exacerbation of an existing disease (a worsening in the character, frequency, or severity of a known condition and recurrence of an intermittent medical condition (e.g., headache) not present at baseline.
Time Frame: From randomization up to Week 12
Population: Safety analysis population included all participants who had received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohorts 1-3: Placebo | Part 2: Cohort 1 and 2 | Part 2: Cohort 3 | Part 2 Cohort 4: Placebo | Part 2: Cohort 4
Number analyzed (Participants) | 6 | 16 | 8 | 5 | 15
percentage of participants | 50.0 | 68.8 | 75.0 | 60.0 | 80.0

4. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of RO7020531 and Its Metabolites Including RO7011785, RO7018822 and RO7033805: SAD and MAD
Time Frame: SAD: Predose and 0.5, 1, 1.5 , 2, 3, 4, 6,8, 12,18, and 24hours post dose on Day 1; MAD: Predose and 0.25, 0.5, 1, 1.5, 2 , 3, 4, 6, 8, 12,18, and 24 hours post dose on Days 1 and 13
Population: The Pharmacokinetic (PK) analysis population included all HVs randomized and adherent to the protocol. Number analyzed is the number of participants available at the specific timepoints.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8 | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
nanograms per milliliter (ng/mL)
  RO7020531: Day 1: number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 0 | 0 | 1
  RO7020531: Day 1 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) |  |  | 1.87 (NA) — Since only 1 participant is analyzed, Standard deviation (SD) was not calculated.
  RO7020531: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RO7011785: Day 1 | 30.2 (10.4) | 115 (69.0) | 182 (71.4) | 508 (203) | 598 (218) | 1270 (505) | 1830 (238) | 1670 (654) | 1060 (428) | 1680 (735) | 2150 (746)
  RO7011785: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7
  RO7011785: Day 13 |  |  |  |  |  |  |  |  | 1100 (448) | 1470 (557) | 2100 (838)
  RO7018822: Day 1 | 2.01 (1.12) | 8.96 (5.15) | 20.0 (16.0) | 52.3 (24.9) | 54.4 (32.1) | 101 (37.7) | 166 (79.3) | 189 (52.5) | 98.3 (42.3) | 144 (52.1) | 234 (163)
  RO7018822: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7
  RO7018822: Day 13 |  |  |  |  |  |  |  |  | 77.7 (42.2) | 125 (47.6) | 220 (143)
  RO7033805: Day 1: number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 1 | 0 | 2
  RO7033805: Day 1 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.285 (0.806) | 1.24 (NA) — Since only 1 participant is analyzed, SD was not calculated. |  | 2.30 (0.339)
  RO7033805: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  RO7033805: Day 13 |  |  |  |  |  |  |  |  |  |  | 1.90 (0.600)

5. Secondary Outcome: Part 2: Cmax of RO7020531 and Its Metabolites Including RO7011785, RO7018822 and RO7033805
Time Frame: Predose and 0.25, 1, 2, 4, 6, 8, and 24 hours post dose on Days 1 and 41
Population: The PK analysis population included all participants randomized and adherent to the protocol. Number analyzed is the number of participants available at the specific timepoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 2: Cohort 3: Participants received RO7020531, 170 mg, along with NUC treatment, orally on Day 1 and QOD for 41 days.
Arm/Group | Part 2: Cohort 1 and 2 | Part 2: Cohort 4 | Part 2: Cohort 3
Number analyzed (Participants) | 16 | 15 | 8
ng/mL
  RO7020531: Day 1: number analyzed (Participants) | 1 | 0 | 0
  RO7020531: Day 1 | 1.70 (NA) — Since only 1 participant is analyzed, SD was not calculated. |  |
  RO7020531: Day 41: number analyzed (Participants) | 0 | 0 | 0
  RO7011785: Day 1 | 1690 (639) | 1500 (668) | 1980 (891)
  RO7011785: Day 41: number analyzed (Participants) | 14 | 12 | 7
  RO7011785: Day 41 | 1580 (591) | 1430 (457) | 1990 (999)
  RO7018822: Day 1 | 167 (93.2) | 203 (110) | 218 (113)
  RO7018822: Day 41: number analyzed (Participants) | 14 | 12 | 7
  RO7018822: Day 41 | 193 (114) | 194 (134) | 184 (90.9)
  RO7033805: Day 1: number analyzed (Participants) | 0 | 1 | 0
  RO7033805: Day 1 |  | 1.43 (NA) — Since only 1 participant is analyzed, SD was not calculated. |
  RO7033805: Day 41: number analyzed (Participants) | 1 | 0 | 0
  RO7033805: Day 41 | 1.51 (NA) — Since only 1 participant is analyzed, SD was not calculated. |  |

6. Secondary Outcome: Part 1: Time to Maximum Observed Plasma Concentration (Tmax) of RO7020531 and Its Metabolites Including RO7011785, RO7018822 and RO7033805: SAD and MAD
Time Frame: as for outcome 4
Population: The PK analysis population included all HVs randomized and adherent to the protocol. Number analyzed is the number of participants available at the specific timepoints.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8 | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
hours (hr)
  RO7020531: Day 1: number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 0 | 0 | 1
  RO7020531: Day 1 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] |  |  | 0.25 [0.25 to 0.25]
  RO7020531: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RO7011785: Day 1 | 0.75 [0.50 to 3.00] | 0.51 [0.50 to 1.50] | 1.00 [0.50 to 1.00] | 0.78 [0.50 to 1.08] | 0.75 [0.50 to 1.00] | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 1.50] | 0.52 [0.50 to 1.50] | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 1.52] | 0.76 [0.50 to 1.00]
  RO7011785: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7
  RO7011785: Day 13 |  |  |  |  |  |  |  |  | 1.00 [0.50 to 1.00] | 1.00 [0.50 to 1.50] | 0.50 [0.50 to 1.50]
  RO7018822: Day 1: number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7
  RO7018822: Day 1 | 0.50 [0.00 to 1.50] | 0.50 [0.50 to 1.50] | 0.50 [0.25 to 1.00] | 0.50 [0.50 to 1.50] | 0.50 [0.50 to 2.00] | 1.00 [0.50 to 2.00] | 0.75 [0.25 to 1.50] | 0.77 [0.50 to 2.00] | 0.75 [0.50 to 2.00] | 1.00 [0.50 to 1.52] | 0.52 [0.50 to 1.00]
  RO7018822: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8
  RO7018822: Day 13 |  |  |  |  |  |  |  |  | 1.00 [0.25 to 2.00] | 0.73 [0.50 to 1.00] | 0.50 [0.50 to 1.00]
  RO7033805: Day 1: number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 1 | 0 | 2
  RO7033805: Day 1 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.50 [0.50 to 0.50] |  | 0.51 [0.50 to 0.52]
  RO7033805: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  RO7033805: Day 13 |  |  |  |  |  |  |  |  |  |  | 0.50 [0.50 to 0.50]

7. Secondary Outcome: Part 2: Tmax of RO7020531 and Its Metabolites Including RO7011785, RO7018822 and RO7033805
Time Frame: Predose and 0.25, 1, 2, 4, 6, 8, and 24 hours post dose on Days 1 and 41
Population: as for outcome 5
Measure: Median (Full Range); unit: hr
Arm/Group | Part 2: Cohort 1 and 2 | Part 2: Cohort 4 | Part 2: Cohort 3
Number analyzed (Participants) | 16 | 15 | 8
hr
  RO7020531: Day 1: number analyzed (Participants) | 1 | 0 | 0
  RO7020531: Day 1 | 0.25 [0.25 to 0.25] |  |
  RO7020531: Day 41: number analyzed (Participants) | 0 | 0 | 0
  RO7011785: Day 1 | 1.00 [0.25 to 2.00] | 1.00 [0.25 to 2.00] | 1.00 [0.92 to 2.00]
  RO7011785: Day 41: number analyzed (Participants) | 14 | 12 | 7
  RO7011785: Day 41 | 1.040 [0.92 to 2.00] | 1.00 [0.92 to 2.00] | 1.00 [0.92 to 4.00]
  RO7018822: Day 1 | 1.00 [0.25 to 2.00] | 1.00 [0.25 to 2.00] | 1.00 [0.25 to 2.00]
  RO7018822: Day 41: number analyzed (Participants) | 14 | 12 | 7
  RO7018822: Day 41 | 1.00 [0.92 to 2.00] | 1.00 [0.25 to 2.00] | 1.00 [0.28 to 4.00]
  RO7033805: Day 1: number analyzed (Participants) | 0 | 1 | 0
  RO7033805: Day 1 |  | 0.25 [0.25 to 0.25] |
  RO7033805: Day 41: number analyzed (Participants) | 1 | 0 | 0
  RO7033805: Day 41 | 1.00 [1.00 to 1.00] |  |

8. Secondary Outcome: Part 1: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUCinf) of RO7020531 and Its Metabolites Including RO7011785, RO7018822 and RO7033805: SAD and MAD
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8 | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
hours*nanogram per milliliter (h*ng/mL)
  RO7020531: Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RO7020531: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RO7011785: Day 1 | 50.9 (28.9) | 138 (40.8) | 253 (58.3) | 596 (103) | 770 (113) | 1600 (228) | 2190 (532) | 2690 (857) | 1450 (278) | 2250 (838) | 2700 (572)
  RO7011785: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7
  RO7011785: Day 13 |  |  |  |  |  |  |  |  | 1420 (288) | 2150 (734) | 2730 (472)
  RO7018822: Day 1: number analyzed (Participants) | 0 | 3 | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 8 | 8
  RO7018822: Day 1 |  | 8.59 (2.61) | 19.0 (5.66) | 43.3 (15.5) | 49.1 (19.9) | 95.4 (21.3) | 139 (40.2) | 224 (81.6) | 97.4 (32.2) | 164 (53.6) | 231 (110)
  RO7018822: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 8 | 6
  RO7018822: Day 13 |  |  |  |  |  |  |  |  | 84.5 (24.0) | 158 (42.1) | 216 (71.4)
  RO7033805: Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RO7033805: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Part 2: AUCinf of RO7020531 and Its Metabolites Including RO7011785, RO7018822 and RO7033805
Time Frame: Predose and 0.25, 1, 2, 4, 6, 8, and 24 hours post dose on Days 1 and 41
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2: Cohort 1 and 2 | Part 2: Cohort 4 | Part 2: Cohort 3
Number analyzed (Participants) | 16 | 15 | 8
h*ng/mL
  RO7020531: Day 1: number analyzed (Participants) | 0 | 0 | 0
  RO7020531: Day 41: number analyzed (Participants) | 0 | 0 | 0
  RO7011785: Day 1: number analyzed (Participants) | 15 | 15 | 8
  RO7011785: Day 1 | 2770 (968) | 2430 (765) | 3060 (1030)
  RO7011785: Day 41: number analyzed (Participants) | 14 | 12 | 7
  RO7011785: Day 41 | 2740 (762) | 2500 (655) | 2960 (909)
  RO7018822: Day 1: number analyzed (Participants) | 5 | 5 | 2
  RO7018822: Day 1 | 338 (147) | 326 (139) | 374 (261)
  RO7018822: Day 41: number analyzed (Participants) | 6 | 5 | 2
  RO7018822: Day 41 | 498 (176) | 482 (249) | 327 (105)
  RO7033805: Day 1: number analyzed (Participants) | 0 | 0 | 0
  RO7033805: Day 41: number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Part 1: Area Under the Plasma Concentration Versus Time Curve up to the Last Measurable Concentration (AUClast) of RO7020531 and Its Metabolites Including RO7011785, RO7018822 and RO7033805: SAD and MAD
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8 | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
h*ng/mL
  RO7020531: Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  RO7020531: Day 1 |  |  |  |  |  |  |  |  |  |  | 0.234 (NA) — Since only 1 participant is analyzed, SD was not calculated.
  RO7020531: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RO7011785: Day 1 | 48.2 (27.3) | 135 (40.1) | 249 (58.8) | 587 (104) | 763 (114) | 1590 (227) | 2180 (533) | 2680 (857) | 1440 (276) | 2240 (837) | 2690 (573)
  RO7011785: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7
  RO7011785: Day 13 |  |  |  |  |  |  |  |  | 1410 (288) | 2150 (733) | 2720 (472)
  RO7018822: Day 1: number analyzed (Participants) | 7 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
  RO7018822: Day 1 | 1.43 (1.47) | 6.73 (2.81) | 16.4 (5.96) | 41.6 (15.5) | 48.5 (19.1) | 93.8 (21.7) | 143 (41.2) | 222 (81.6) | 95.9 (32.3) | 161 (52.9) | 228 (109)
  RO7018822: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7
  RO7018822: Day 13 |  |  |  |  |  |  |  |  | 80.6 (23.5) | 154 (39.7) | 210 (64.9)
  RO7033805: Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  RO7033805: Day 1 |  |  |  |  |  |  |  | 0.285 (NA) — Since only 1 participant is analyzed, SD was not calculated. | 0.155 (NA) — Since only 1 participant is analyzed, SD was not calculated. |  | 0.434 (0.224)
  RO7033805: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  RO7033805: Day 13 |  |  |  |  |  |  |  |  |  |  | 0.316 (0.155)

11. Secondary Outcome: Part 2: AUClast of RO7020531 and Its Metabolites Including RO7011785, RO7018822 and RO7033805
Time Frame: Predose and 0.25, 1, 2, 4, 6, 8, and 24 hours post dose on Days 1 and 41
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2: Cohort 1 and 2 | Part 2: Cohort 4 | Part 2: Cohort 3
Number analyzed (Participants) | 16 | 15 | 8
h*ng/mL
  RO7020531: Day 1: number analyzed (Participants) | 1 | 0 | 0
  RO7020531: Day 1 | 0.213 (NA) — Since only 1 participant is analyzed, SD was not calculated. |  |
  RO7020531: Day 41: number analyzed (Participants) | 0 | 0 | 0
  RO7011785: Day 1 | 2820 (979) | 2400 (762) | 3030 (1040)
  RO7011785: Day 41: number analyzed (Participants) | 14 | 12 | 7
  RO7011785: Day 41 | 2730 (771) | 2470 (653) | 2930 (915)
  RO7018822: Day 1 | 220 (124) | 253 (127) | 255 (134)
  RO7018822: Day 41: number analyzed (Participants) | 14 | 12 | 7
  RO7018822: Day 41 | 297 (214) | 301 (228) | 243 (87.8)
  RO7033805: Day 1: number analyzed (Participants) | 0 | 1 | 0
  RO7033805: Day 1 |  | 0.179 (NA) — Since only 1 participant is analyzed, SD was not calculated. |
  RO7033805: Day 41: number analyzed (Participants) | 1 | 0 | 0
  RO7033805: Day 41 | 0.566 (NA) — Since only 1 participant is analyzed, SD was not calculated. |  |

12. Secondary Outcome: Part 1: Half Life (t1/2) of RO7020531 and Its Metabolites Including RO7011785, RO7018822 and RO7033805: SAD and MAD
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8 | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
hr
  RO7020531: Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RO7020531: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RO7011785: Day 1 | 1.11 (0.370) | 1.56 (0.319) | 1.81 (0.506) | 2.78 (0.479) | 2.82 (0.599) | 3.35 (0.573) | 3.26 (0.254) | 3.39 (0.616) | 3.23 (0.635) | 2.80 (0.538) | 3.00 (0.692)
  RO7011785: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7
  RO7011785: Day 13 |  |  |  |  |  |  |  |  | 3.63 (0.740) | 3.23 (0.528) | 3.45 (1.12)
  RO7018822: Day 1: number analyzed (Participants) | 0 | 3 | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 8 | 8
  RO7018822: Day 1 |  | 0.610 (0.0986) | 0.655 (0.276) | 0.579 (0.144) | 0.567 (0.190) | 0.585 (0.0780) | 0.564 (0.0827) | 0.645 (0.137) | 0.548 (0.111) | 0.586 (0.0507) | 0.601 (0.113)
  RO7018822: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 8 | 6
  RO7018822: Day 13 |  |  |  |  |  |  |  |  | 0.578 (0.0528) | 0.620 (0.0812) | 0.744 (0.204)
  RO7033805: Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RO7033805: Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Part 2: t1/2 of RO7020531 and Its Metabolites Including RO7011785, RO7018822 and RO7033805
Time Frame: Predose and 0.25, 1, 2, 4, 6, 8, and 24 hours post dose on Days 1 and 41
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 2: Cohort 1 and 2 | Part 2: Cohort 4 | Part 2: Cohort 3
Number analyzed (Participants) | 16 | 15 | 8
hr
  RO7020531: Day 1: number analyzed (Participants) | 0 | 0 | 0
  RO7020531: Day 41: number analyzed (Participants) | 0 | 0 | 0
  RO7011785: Day 1: number analyzed (Participants) | 15 | 15 | 8
  RO7011785: Day 1 | 3.09 (0.982) | 2.63 (1.19) | 3.06 (0.934)
  RO7011785: Day 41: number analyzed (Participants) | 14 | 12 | 7
  RO7011785: Day 41 | 3.09 (0.697) | 2.77 (1.19) | 2.90 (0.980)
  RO7018822: Day 1: number analyzed (Participants) | 5 | 5 | 2
  RO7018822: Day 1 | 1.19 (0.886) | 0.665 (0.0431) | 0.648 (0.0317)
  RO7018822: Day 41: number analyzed (Participants) | 6 | 5 | 2
  RO7018822: Day 41 | 0.776 (0.146) | 0.714 (0.112) | 0.720 (0.774)
  RO7033805: Day 1: number analyzed (Participants) | 0 | 0 | 0
  RO7033805: Day 41: number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Part 1: Total Amount of RO7020531, RO7011785, RO7018822 and RO7033805 in Urine: SAD
Description: Total amount of the study drug and metabolites recovered in urine was reported.
Time Frame: 0 to 24 hrs Postdose on Day 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
mg
  RO7020531: number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 5 | 0
  RO7020531 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) |
  RO7011785 | 1.70 (0.274) | 5.04 (1.23) | 11.0 (1.92) | 18.2 (8.96) | 25.5 (7.81) | 48.1 (17.7) | 68.6 (16.7) | 83.5 (17.4)
  RO7018822 | 0.0137 (0.0167) | 0.0754 (0.0274) | 0.188 (0.0399) | 0.271 (0.171) | 0.372 (0.145) | 0.728 (0.337) | 1.10 (0.417) | 1.87 (1.00)
  RO7033805: number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 5 | 0
  RO7033805 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) |

15. Secondary Outcome: Part 1:Mean Concentration of Interferon Alpha (IFN-alpha): SAD and MAD
Description: Mean concentrations of IFN-alpha for SAD were calculated following single-dose and for MAD it was calculated following multiple doses. The standard deviation (SD) presented is actually the log transformed geometric standard deviation.
Time Frame: SAD: Predose, 2, 6, 12 and 24 hrs Postdose; MAD: Predose, 2, 6, 12, and 24 hrs Postdose on Day 1; Predose, 2, 6 and 24 hrs Postdose on Days 3, 5, 7, 13 and 20
Population: Pharmacodynamic population included all HVs who had received at least 1 dose of the study drug and with PD data available.
Measure: Geometric Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Part 1 Cohorts 1-8 SAD: Placebo | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8 | Part 1 Cohorts 1-3, MAD: Placebo | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 8 | 8
picogram per milliliter (pg/mL) | 0.0484 (1.3166) | 0.0475 (1.4288) | 0.0438 (1.1316) | 0.0447 (1.1166) | 0.0436 (1.0600) | 0.0494 (1.5718) | 0.0533 (1.5205) | 0.1385 (3.8417) | 0.1358 (3.8126) | 0.0530 (1.0135) | 0.0761 (1.9769) | 0.1148 (3.1080) | 0.3349 (5.5985)

16. Secondary Outcome: Part 2: Mean Concentration of IFN-alpha
Description: Mean concentrations of IFN-alpha for Part 2 were calculated following multiple doses. The SD presented is actually the log transformed geometric standard deviation.
Time Frame: Predose, 6, 8 and 24 hrs Postdose on Day 1; Predose, 4-6, 24 hrs Postdose on Days 3, 7 and 21; Predose, 6, 24 hrs Postdose on Day 41
Population: Pharmacodynamic population included all participants who had received at least 1 dose of the study drug and with PD data available.
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Groups:
- Part 2 Cohort 3: Participants received RO7020531, 170 mg, along with NUC treatment, orally, on Day 1 and QOD for 41 days.
Arm/Group | Part 2 Cohorts 1-3: Placebo | Part 2: Cohort 1 and 2 | Part 2 Cohort 3 | Part 2 Cohort 4: Placebo | Part 2: Cohort 4
Number analyzed (Participants) | 6 | 16 | 8 | 5 | 15
pg/mL | 0.0533 (1.0668) | 0.3801 (9.1442) | 0.2831 (9.0521) | 0.0574 (1.2737) | 0.3161 (8.0853)

17. Secondary Outcome: Part 1: Mean Fold Change From Baseline in Cytokine Markers: SAD and MAD
Description: Cytokines markers include Chemokine (C-X-C Motif) Ligand 10 (IP-10), Interleukin 6 (IL-6), Interleukin 10 (IL-10), Interleukin 12 p40 (IL-12 p40), Neopterin, Tumor Necrosis Factor-Alpha (TNF-alpha). The SD presented is actually the log transformed geometric standard deviation.
Time Frame: SAD: Predose, 2, 6, 12, 24, 48 (only Neopterin) and 96 hrs (only Neopterin) Postdose; MAD: Predose, 2, 6, 12, and 24 hrs Postdose on Day 1; Predose, 2, 6 and 24 hrs Postdose on Days 3, 5, 7, 13 and 20
Population: as for outcome 15
Measure: Geometric Mean (Standard Deviation); unit: Fold change
Arm/Group | Part 1 Cohorts 1-8 SAD: Placebo | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8 | Part 1 Cohorts 1-3, MAD: Placebo | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 8 | 8
Fold change
  Neopterin | 0.9861 (1.1833) | 1.0561 (1.3678) | 1.0175 (1.2665) | 0.9878 (1.2300) | 0.9975 (1.1503) | 0.9896 (1.2475) | 0.9738 (1.1791) | 1.0688 (1.3926) | 1.1257 (1.4298) | 0.9331 (1.1446) | 1.5842 (1.3637) | 1.1228 (1.5260) | 1.5453 (1.5431)
  IP-10 | 0.9067 (1.3101) | 0.8751 (1.4713) | 0.9112 (1.3624) | 0.9250 (1.2966) | 0.9754 (1.2328) | 0.9267 (1.2754) | 1.0390 (1.2198) | 1.6532 (2.0266) | 1.2909 (1.8003) | 1.0256 (1.4853) | 1.2010 (1.4186) | 1.2076 (1.7543) | 1.7327 (2.3938)
  IL-12 p40 | 1.0276 (1.2232) | 0.9414 (1.3431) | 1.0419 (1.2198) | 0.9706 (1.0957) | 1.0000 (1.0000) | 1.0012 (1.0156) | 1.0000 (1.0000) | 1.0025 (1.1817) | 1.0009 (1.0049) | 0.6782 (1.7025) | 0.8672 (1.3474) | 0.9588 (1.3470) | 0.9002 (1.3373)
  IL-10 | 0.9692 (1.5013) | 0.7042 (2.0970) | 1.0568 (1.5139) | 0.9622 (1.3461) | 0.9483 (1.4871) | 0.7451 (2.3095) | 1.0047 (1.3322) | 1.1900 (1.6328) | 1.1926 (1.4208) | 0.6841 (3.4286) | 1.0961 (1.4560) | 0.8834 (1.5662) | 1.1232 (1.5901)
  IL-6 | 1.4493 (2.4225) | 1.9626 (2.9840) | 1.2293 (1.9209) | 1.2464 (2.5694) | 1.2857 (1.8437) | 0.9486 (1.9942) | 1.3207 (2.0960) | 1.4167 (2.3111) | 1.6928 (2.1981) | 1.8290 (2.8323) | 1.3521 (2.2473) | 1.9065 (2.2325) | 1.1306 (2.3792)
  TNF-alpha | 1.0875 (1.8701) | 1.0374 (1.7561) | 0.9435 (1.4360) | 0.8698 (2.1721) | 1.0781 (1.4358) | 0.8825 (1.7991) | 0.9249 (1.6530) | 0.9663 (1.7846) | 1.1756 (1.5505) | 1.0830 (1.6154) | 1.2136 (1.5828) | 0.9887 (1.5106) | 0.8985 (1.6625)

18. Secondary Outcome: Part 2: Mean Fold Change From Baseline in Cytokine Markers
Description: Cytokines markers included IP- 10, IL- 6, IL-1 10, IL-12 p40, Neopterin and TNF -alpha. The SD presented is actually the log transformed geometric standard deviation.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Geometric Mean (Standard Deviation); unit: Fold change
Arm/Group | Part 2 Cohorts 1-3: Placebo | Part 2: Cohort 1 and 2 | Part 2 Cohort 3 | Part 2 Cohort 4: Placebo | Part 2: Cohort 4
Number analyzed (Participants) | 6 | 16 | 8 | 5 | 15
Fold change
  Neopterin | 1.0473 (1.2426) | 1.5596 (1.7824) | 1.7935 (1.9267) | 1.0591 (1.5154) | 1.4676 (1.7203)
  IP-10 | 0.9007 (1.3368) | 2.2323 (2.6810) | 2.1018 (2.9560) | 0.8939 (1.3557) | 1.8598 (2.6359)
  IL-12 p40 | 1.0000 (1.0000) | 1.0109 (1.1763) | 0.9624 (1.1261) | 1.0000 (1.0000) | 0.9740 (1.1886)
  IL-10 | 1.0428 (1.3767) | 1.2587 (1.5415) | 1.3441 (1.9726) | 0.8232 (1.6060) | 1.2540 (1.8818)
  IL-6 | 1.0172 (1.1251) | 1.0909 (1.4962) | 1.4235 (2.1969) | 0.8127 (1.4478) | 1.1596 (1.6084)
  TNF-alpha | 0.9848 (1.4186) | 1.2674 (1.6169) | 1.0527 (1.6605) | 1.0415 (1.3014) | 1.0418 (1.5470)

19. Secondary Outcome: Part 1:Mean Fold Change From Baseline in Markers of Transcriptional Responses: SAD and MAD
Description: Markers of transcriptional responses includes messenger ribonucleic acid interferon-stimulated gene 15(mRNA ISG15), messenger RNA oligoadenylate synthetase 1 (mRNA OAS1), messenger RNA myxovirus resistance 1 gene (mRNA MX-1), messenger RNA Toll-like receptor (mRNA TLR7). The SD presented is actually the log transformed geometric standard deviation.
Time Frame: SAD: Predose, 2, 6, 12 and 24 Postdose; MAD: Predose, 2, 6, 12, and 24 hrs Postdose on Day 1; Predose, 2, 6 and 24 hrs Postdose on Days 3, 5, 7, 13 and 20
Population: as for outcome 15
Measure: Geometric Mean (Standard Deviation); unit: Fold change
Arm/Group | Part 1 Cohorts 1-8 SAD: Placebo | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8 | Part 1 Cohorts 1-3, MAD: Placebo | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 8 | 8
Fold change
  mRNA ISG15 | 0.9709 (1.2752) | 1.1708 (1.9326) | 1.0525 (1.3985) | 0.9386 (1.5924) | 1.0799 (1.3980) | 1.0190 (1.6295) | 1.6951 (2.5735) | 3.0359 (4.0456) | 3.1083 (3.9014) | 1.1703 (1.6841) | 1.9408 (2.6372) | 2.3632 (2.8453) | 4.8748 (4.1091)
  mRNA OAS1 | 1.0251 (1.2295) | 1.0414 (1.4571) | 1.0338 (1.2876) | 0.9666 (1.4060) | 0.8584 (1.7499) | 1.0680 (1.4851) | 1.4093 (1.7808) | 2.3437 (2.5254) | 2.2308 (2.4993) | 1.0651 (1.5253) | 1.8186 (2.3871) | 2.1467 (2.2610) | 3.2312 (3.0239)
  mRNA Mx-1 | 1.0179 (1.3078) | 0.9750 (1.5209) | 1.0166 (1.4143) | 0.9045 (1.4844) | 0.8811 (1.5884) | 1.0837 (1.6314) | 1.5271 (2.3070) | 2.8672 (3.5170) | 2.6646 (3.0944) | 0.9813 (1.5661) | 2.3613 (2.8339) | 2.0847 (2.8118) | 3.2388 (3.9277)
  mRNA TLR7 | 1.0698 (1.3124) | 1.1518 (1.3697) | 1.0401 (1.2667) | 1.0658 (1.2237) | 1.0965 (1.3698) | 1.1289 (1.2710) | 1.2120 (1.3328) | 1.5925 (1.6473) | 1.5596 (2.1403) | 1.2315 (1.6428) | 1.2089 (1.6716) | 1.2626 (1.5696) | 1.6081 (1.8082)

20. Secondary Outcome: Part 2: Mean Fold Change From Baseline in Markers of Transcriptional Responses
Description: Transcriptional markers include mRNA ISG15, mRNA OAS1, mRNA MX-1, mRNA TLR7. The SD presented is actually the log transformed geometric standard deviation.
Time Frame: Predose, 6, 8, 24 hrs postdose on Day 1; Predose, 4-6, 24 hrs postdose on Days 3, 7, 21; Predose, 6, 24 hrs postdose on Day 41
Population: as for outcome 16
Measure: Geometric Mean (Standard Deviation); unit: Fold change
Arm/Group | Part 2 Cohorts 1-3: Placebo | Part 2: Cohort 1 and 2 | Part 2 Cohort 3 | Part 2 Cohort 4: Placebo | Part 2: Cohort 4
Number analyzed (Participants) | 6 | 16 | 8 | 5 | 15
Fold change
  mRNA ISG15 | 1.0745 (1.6135) | 4.2007 (3.9059) | 6.8997 (4.1313) | 0.8661 (1.5914) | 3.9424 (3.3660)
  mRNA OAS1 | 0.9617 (1.2926) | 3.1021 (2.6766) | 4.0466 (2.7318) | 0.7973 (1.4425) | 3.0355 (2.4692)
  mRNA Mx-1 | 0.9140 (1.4847) | 3.1760 (3.2606) | 5.0962 (3.3744) | 0.8296 (1.3309) | 3.4811 (2.9921)
  mRNA TLR7 | 1.0848 (1.4306) | 1.5280 (1.7527) | 1.5745 (1.7411) | 1.0240 (1.3620) | 1.3211 (1.9422)

21. Secondary Outcome: Effect of RO7020531 Dosing on ECG Parameters (PR [PQ], QRS, QT, QTcF in Miliseconds [ms]) Using Exposure-response Analysis: SAD and MAD
Time Frame: SAD: Predose, 0.5, 1, 2, 4, 6, 12, 24 and 48 hrs Post dose on Day 1; MAD: Predose, 0.5, 1,2,4 and 12 hrs Postdose on Day 1 and 13; Predose, 2 and 6 hrs Postdose on Day 3, Predose, 6 and 24 hrs Postdose on Day , 7, 9, and 11
Population: Data was not collected for this Outcome Measure due to change in planned analyses. This analysis will be performed after CSR finalization, as its results will only be required before executing a Phase 3 study with RO7020531.
Arm/Group | Part 1 Cohorts 1-8 SAD: Placebo | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8 | Part 1 Cohorts 1-3, MAD: Placebo | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Part 2: Plasma Concentrations of Tenofovir, Tenofovir Alafenamide, Entecavir, Adefovir and Telbivudine
Description: Adefovir was not administered to any participants in the study. Hence, no data could be collected for plasma concentration of adefovir. As participants in each cohort received different NUCs the data for Cohorts 1, 2 and 3 have been reported separately.
Time Frame: Pre-dose and 2-4 hours post-dose on Day 1, Day 21 and Day 41
Population: The PK analysis population included all participants randomised and adherent to the protocol. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants available at the specific timepoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 2 Cohorts 1: Participants received RO7020531, 150 mg, along with NUC treatment, orally, on Day 1 and QOD for 41 days.
- Part 2 Cohort 2: Participants were enrolled in Cohort 2 after the internal monitoring committee (IMC) assessed the safety and tolerability data available for Cohort 1. Participants received RO7020531, 150 mg, along with NUC treatment, orally, on Day 1 and QOD for 41 days.
- Part 2 Cohort 3: Participants received RO7020531, 170 mg, along with NUC treatment , orally QOD from Day 1 through to Day 41.
Arm/Group | Part 2 Cohorts 1 | Part 2 Cohort 2 | Part 2 Cohort 3
Number analyzed (Participants) | 6 | 5 | 5
ng/mL
  Entecavir - Day 1: Predose: number analyzed (Participants) | 4 | 4 | 5
  Entecavir - Day 1: Predose | 0.467 (0.13) | 0.420 (0.10) | 0.590 (0.62)
  Entecavir - Day 1: 2-4 hours Post Dose: number analyzed (Participants) | 4 | 4 | 5
  Entecavir - Day 1: 2-4 hours Post Dose | 1.974 (1.08) | 1.455 (0.53) | 1.019 (0.60)
  Entecavir - Day 21: Predose: number analyzed (Participants) | 4 | 3 | 4
  Entecavir - Day 21: Predose | 0.494 (0.07) | 0.365 (0.09) | 0.810 (0.92)
  Entecavir - Day 21: 2-4 hours Post Dose: number analyzed (Participants) | 4 | 4 | 4
  Entecavir - Day 21: 2-4 hours Post Dose | 1.543 (0.76) | 1.568 (0.80) | 0.935 (0.20)
  Entecavir - Day 41: Predose: number analyzed (Participants) | 3 | 4 | 3
  Entecavir - Day 41: Predose | 0.406 (0.10) | 0.308 (0.08) | 0.887 (0.89)
  Entecavir - Day 41: 2-4 hours Post Dose: number analyzed (Participants) | 3 | 4 | 4
  Entecavir - Day 41: 2-4 hours Post Dose | 1.373 (0.66) | 1.267 (0.50) | 1.427 (0.69)
  Tenofovir - Day 1: Predose | 54.93 (32.7) | 60.00 (26.5) | 71.12 (35.7)
  Tenofovir - Day 1: 2-4 hours Post Dose | 155.1 (106) | 214.2 (64.0) | 245.0 (49.8)
  Tenofovir - Day 21: Predose: number analyzed (Participants) | 5 | 4 | 5
  Tenofovir - Day 21: Predose | 63.90 (29.5) | 58.40 (21.4) | 57.02 (28.0)
  Tenofovir - Day 21: 2-4 hours Post Dose: number analyzed (Participants) | 5 | 5 | 5
  Tenofovir - Day 21: 2-4 hours Post Dose | 206.6 (81.4) | 273.0 (177) | 222.2 (70.8)
  Tenofovir - Day 41: Predose: number analyzed (Participants) | 5 | 5 | 5
  Tenofovir - Day 41: Predose | 66.82 (34.0) | 64.06 (32.7) | 56.56 (26.3)
  Tenofovir - Day 41: 2-4 hours Post Dose: number analyzed (Participants) | 5 | 5 | 5
  Tenofovir - Day 41: 2-4 hours Post Dose | 250.9 (108) | 250.4 (112) | 188.4 (58.7)
  Tenofovir Alafenamide - Day 1: Predose: number analyzed (Participants) | 0 | 0 | 0
  Tenofovir Alafenamide - Day 1: 2-4 hours Post Dose: number analyzed (Participants) | 0 | 1 | 0
  Tenofovir Alafenamide - Day 1: 2-4 hours Post Dose |  | 0.058 (0.058) |
  Tenofovir Alafenamide - Day 21: Predose: number analyzed (Participants) | 0 | 0 | 0
  Tenofovir Alafenamide - Day 21: 2-4 hours Post Dose: number analyzed (Participants) | 0 | 0 | 0
  Tenofovir Alafenamide - Day 41: Predose: number analyzed (Participants) | 0 | 0 | 0
  Tenofovir Alafenamide - Day 41: 2-4 hours Post Dose: number analyzed (Participants) | 0 | 0 | 0
  Telbivudine - Day 1: Predose: number analyzed (Participants) | 0 | 1 | 1
  Telbivudine - Day 1: Predose |  | 602.0 (602.0) | 330.0 (330.0)
  Telbivudine - Day 1: 2-4 hours Post Dose: number analyzed (Participants) | 0 | 1 | 1
  Telbivudine - Day 1: 2-4 hours Post Dose |  | 4760 (4760) | 2820 (2820)
  Telbivudine - Day 21: Predose: number analyzed (Participants) | 0 | 1 | 1
  Telbivudine - Day 21: Predose |  | 1030 (1030) | 314.0 (314.0)
  Telbivudine - Day 21: 2-4 hours Post Dose: number analyzed (Participants) | 0 | 1 | 1
  Telbivudine - Day 21: 2-4 hours Post Dose |  | 2030 (2030) | 1790 (1790)
  Telbivudine - Day 41: Predose: number analyzed (Participants) | 0 | 1 | 1
  Telbivudine - Day 41: Predose |  | 935.0 (935.0) | 260.0 (260.0)
  Telbivudine - Day 41: 2-4 hours Post Dose: number analyzed (Participants) | 0 | 1 | 1
  Telbivudine - Day 41: 2-4 hours Post Dose |  | 2850 (2850) | 2450 (2450)

23. Primary Outcome: Part 1: Percentage of SAD Participants With Laboratory Abnormalities Based on Hematology, Clinical Chemistry, Coagulation and Urinalysis Test Results
Description: For all laboratory parameters included, there exists a Roche predefined standard reference range. Laboratory values falling outside this standard reference range were labeled "H" for high or "L" for low in HV/participant listings of laboratory data.
Time Frame: From randomization up to Day 8
Population: Safety population included all HVs who had received at least 1 dose of study drug. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-8 SAD: Placebo | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
percentage of participants
  Eosinophils Absolute - High: number analyzed (Participants) | 16 | 8 | 8 | 7 | 8 | 7 | 6 | 8 | 8
  Eosinophils Absolute - High | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0
  Erythrocyte Mean Corpuscular HGB Concentration - Low: number analyzed (Participants) | 14 | 6 | 8 | 8 | 8 | 8 | 8 | 8 | 8
  Erythrocyte Mean Corpuscular HGB Concentration - Low | 0 | 0 | 12.5 | 12.5 | 0 | 0 | 12.5 | 0 | 12.5
  Erythrocyte Mean Corpuscular Hemoglobin - Low: number analyzed (Participants) | 15 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
  Erythrocyte Mean Corpuscular Hemoglobin - Low | 6.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocyte Mean Corpuscular Volume - High | 0 | 0 | 12.5 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit - Low: number analyzed (Participants) | 15 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
  Hematocrit - Low | 6.7 | 25.0 | 12.5 | 0 | 0 | 0 | 25.0 | 12.5 | 12.5
  Hemoglobin - Low | 6.3 | 25.0 | 12.5 | 12.5 | 0 | 25.0 | 0 | 25.0 | 0
  Hemoglobin - High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5
  Lymphocytes Absolute - Low | 0 | 12.5 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5
  Monocytes Absolute - High: number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 7 | 8
  Monocytes Absolute - High | 0 | 12.5 | 12.5 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils, Total, Absolute - Low: number analyzed (Participants) | 14 | 7 | 8 | 8 | 8 | 6 | 7 | 8 | 7
  Neutrophils, Total, Absolute - Low | 7.1 | 14.3 | 12.5 | 0 | 0 | 16.7 | 0 | 12.5 | 0
  Neutrophils, Total, Absolute - High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5 | 0
  Platelet - Low: number analyzed (Participants) | 16 | 7 | 8 | 8 | 8 | 8 | 8 | 8 | 8
  Platelet - Low | 0 | 0 | 0 | 0 | 12.5 | 0 | 12.5 | 0 | 0
  Platelet - High: number analyzed (Participants) | 16 | 8 | 8 | 8 | 7 | 8 | 8 | 8 | 8
  Platelet - High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5 | 0
  Red Blood Cell Count - Low: number analyzed (Participants) | 16 | 7 | 8 | 8 | 8 | 8 | 8 | 8 | 7
  Red Blood Cell Count - Low | 6.3 | 0 | 12.5 | 0 | 0 | 12.5 | 12.5 | 0 | 0
  Red Blood Cell Count - High: number analyzed (Participants) | 15 | 8 | 8 | 8 | 8 | 8 | 7 | 8 | 8
  Red Blood Cell Count - High | 6.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reticulocytes, Pct - High | 0 | 0 | 12.5 | 0 | 12.5 | 0 | 0 | 0 | 0
  White Blood Cell Count - Low: number analyzed (Participants) | 15 | 6 | 6 | 8 | 8 | 8 | 7 | 8 | 7
  White Blood Cell Count - Low | 13.3 | 0 | 0 | 12.5 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Count - High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5 | 0
  Albumin - Low: number analyzed (Participants) | 15 | 8 | 7 | 8 | 7 | 8 | 7 | 8 | 8
  Albumin - Low | 0 | 0 | 0 | 0 | 0 | 0 | 14.3 | 12.5 | 12.5
  Alkaline Phosphatase - Low: number analyzed (Participants) | 13 | 7 | 8 | 8 | 8 | 8 | 8 | 8 | 8
  Alkaline Phosphatase - Low | 0 | 0 | 0 | 0 | 0 | 0 | 12.5 | 0 | 0
  Alkaline Phosphatase - High | 0 | 0 | 0 | 12.5 | 0 | 0 | 0 | 0 | 0
  Bicarbonate CO2 - Low: number analyzed (Participants) | 16 | 8 | 8 | 6 | 8 | 8 | 8 | 7 | 8
  Bicarbonate CO2 - Low | 6.3 | 0 | 12.5 | 0 | 12.5 | 0 | 0 | 0 | 12.5
  Blood Glucose, Fasting - High: number analyzed (Participants) | 14 | 8 | 6 | 8 | 8 | 5 | 7 | 8 | 7
  Blood Glucose, Fasting - High | 7.1 | 12.5 | 50.0 | 0 | 0 | 0 | 42.9 | 12.5 | 14.3
  Blood Urea Nitrogen - Low: number analyzed (Participants) | 14 | 8 | 8 | 7 | 7 | 7 | 8 | 5 | 5
  Blood Urea Nitrogen - Low | 7.1 | 12.5 | 0 | 14.3 | 14.3 | 0 | 0 | 40.0 | 40.0
  Blood Urea Nitrogen - High | 6.3 | 0 | 12.5 | 0 | 0 | 0 | 12.5 | 0 | 0
  Calcium - High | 6.3 | 0 | 0 | 0 | 0 | 12.5 | 0 | 0 | 0
  Chloride - Low: number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 8
  Chloride - Low | 6.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5
  Cholesterol - High: number analyzed (Participants) | 12 | 5 | 4 | 8 | 4 | 5 | 6 | 7 | 7
  Cholesterol - High | 8.3 | 20.0 | 0 | 0 | 25.0 | 0 | 16.7 | 14.3 | 0
  Creatinine - Low: number analyzed (Participants) | 15 | 8 | 6 | 8 | 8 | 7 | 8 | 8 | 8
  Creatinine - Low | 0 | 12.5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine - High | 0 | 0 | 12.5 | 0 | 0 | 0 | 12.5 | 0 | 0
  Cystatin C - Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5
  Cystatin C - High: number analyzed (Participants) | 15 | 8 | 8 | 8 | 8 | 7 | 7 | 8 | 8
  Cystatin C - High | 13.3 | 12.5 | 0 | 0 | 12.5 | 0 | 0 | 12.5 | 25.0
  Direct Bilirubin - High: number analyzed (Participants) | 14 | 8 | 7 | 6 | 7 | 6 | 7 | 8 | 8
  Direct Bilirubin - High | 14.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Phosphorus - High | 6.3 | 0 | 0 | 0 | 12.5 | 0 | 0 | 12.5 | 0
  Potassium - Low: number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7
  Potassium - Low | 0 | 0 | 0 | 0 | 12.5 | 0 | 0 | 0 | 0
  Protein, Total - Low: number analyzed (Participants) | 15 | 7 | 8 | 8 | 8 | 8 | 6 | 7 | 8
  Protein, Total - Low | 20.0 | 14.3 | 25.0 | 25.0 | 12.5 | 25.0 | 16.7 | 28.6 | 12.5
  Protein, Total - High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5
  SGOT/AST - High | 0 | 0 | 12.5 | 0 | 0 | 12.5 | 0 | 12.5 | 0
  SGPT/ALT - High: number analyzed (Participants) | 16 | 8 | 8 | 6 | 7 | 8 | 8 | 7 | 8
  SGPT/ALT - High | 0 | 0 | 12.5 | 0 | 14.3 | 12.5 | 0 | 0 | 12.5
  Sodium - High | 6.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Triglycerides, Fasting - High: number analyzed (Participants) | 15 | 7 | 7 | 8 | 7 | 7 | 7 | 7 | 7
  Triglycerides, Fasting - High | 0 | 0 | 14.3 | 0 | 28.6 | 0 | 0 | 0 | 0
  Uric Acid - High: number analyzed (Participants) | 14 | 8 | 8 | 7 | 8 | 7 | 6 | 8 | 7
  Uric Acid - High | 7.1 | 0 | 0 | 14.3 | 25.0 | 0 | 16.7 | 12.5 | 0
  Creatinine Clearance - Low: number analyzed (Participants) | 16 | 7 | 6 | 8 | 8 | 8 | 8 | 8 | 8
  Creatinine Clearance - Low | 0 | 0 | 0 | 0 | 0 | 0 | 35.7 | 0 | 0
  Creatinine Clearance - High: number analyzed (Participants) | 13 | 6 | 6 | 5 | 5 | 4 | 6 | 2 | 6
  Creatinine Clearance - High | 23.1 | 0 | 16.7 | 20.0 | 20.0 | 25.0 | 0 | 0 | 0

24. Primary Outcome: Part 1: Percentage of MAD Participants With Laboratory Abnormalities Based on Hematology, Clinical Chemistry, Coagulation and Urinalysis Test Results
Description: as for outcome 23
Time Frame: From randomization up to Day 20
Population: Safety analysis population included all HVs who had received at least 1 dose of study drug. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-3, MAD: Placebo | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 6 | 8 | 8 | 8
percentage of participants
  Eosinophils Absolute - High: number analyzed (Participants) | 5 | 8 | 8 | 7
  Eosinophils Absolute - High | 0 | 12.5 | 0 | 0
  Erythrocyte Mean Corpuscular HGB Concentration - Low: number analyzed (Participants) | 6 | 8 | 7 | 7
  Erythrocyte Mean Corpuscular HGB Concentration - Low | 0 | 0 | 28.6 | 42.9
  Erythrocyte Mean Corpuscular HGB Concentration - High: number analyzed (Participants) | 6 | 7 | 8 | 8
  Erythrocyte Mean Corpuscular HGB Concentration - High | 0 | 14.3 | 0 | 0
  Erythrocyte Mean Corpuscular Hemoglobin - Low: number analyzed (Participants) | 6 | 7 | 8 | 8
  Erythrocyte Mean Corpuscular Hemoglobin - Low | 0 | 0 | 0 | 12.5
  Hematocrit - Low | 16.7 | 62.5 | 62.5 | 37.5
  Hemoglobin - Low | 16.7 | 50.0 | 62.5 | 37.5
  Neutrophils, Total, Absolute: number analyzed (Participants) | 6 | 8 | 6 | 8
  Neutrophils, Total, Absolute | 16.7 | 25.0 | 16.7 | 37.5
  Red blood cell count - Low | 0 | 0 | 25.0 | 25.0
  Reticulocytes, Pct - High: number analyzed (Participants) | 5 | 8 | 8 | 8
  Reticulocytes, Pct - High | 0 | 0 | 25.0 | 12.5
  White Blood Cell Count - Low: number analyzed (Participants) | 5 | 8 | 5 | 8
  White Blood Cell Count - Low | 0 | 0 | 20.0 | 25.0
  Albumin - Low: number analyzed (Participants) | 5 | 8 | 8 | 8
  Albumin - Low | 40.0 | 37.5 | 37.5 | 25.0
  Alkaline Phosphatase - Low: number analyzed (Participants) | 6 | 7 | 8 | 7
  Alkaline Phosphatase - Low | 0 | 0 | 12.5 | 0
  Bicarbonate CO2 - Low: number analyzed (Participants) | 6 | 8 | 7 | 8
  Bicarbonate CO2 - Low | 16.7 | 12.5 | 0 | 0
  Blood Glucose, Fasting - High: number analyzed (Participants) | 5 | 8 | 6 | 7
  Blood Glucose, Fasting - High | 20.0 | 12.5 | 16.7 | 14.3
  Blood Urea Nitrogen - Low: number analyzed (Participants) | 6 | 6 | 5 | 4
  Blood Urea Nitrogen - Low | 33.3 | 33.3 | 80.0 | 100.0
  Cholesterol - High: number analyzed (Participants) | 6 | 8 | 5 | 7
  Cholesterol - High | 16.7 | 12.5 | 20.0 | 14.3
  Creatinine - Low: number analyzed (Participants) | 6 | 8 | 8 | 7
  Creatinine - Low | 0 | 25.0 | 0 | 42.9
  Cystatin C - High: number analyzed (Participants) | 6 | 6 | 8 | 8
  Cystatin C - High | 0 | 33.3 | 0 | 0
  Direct Bilirubin - High: number analyzed (Participants) | 5 | 7 | 7 | 7
  Direct Bilirubin - High | 20.0 | 14.3 | 0 | 14.3
  Phosphorus - High | 0 | 12.5 | 12.5 | 25.0
  Protein, Total - Low: number analyzed (Participants) | 4 | 8 | 8 | 8
  Protein, Total - Low | 25.0 | 75.0 | 50.0 | 62.5
  SGOT/AST - High | 0 | 12.5 | 0 | 0
  SGPT/ALT - High: number analyzed (Participants) | 6 | 8 | 8 | 7
  SGPT/ALT - High | 0 | 12.5 | 0 | 14.3
  Uric Acid - Low | 0 | 12.5 | 0 | 0
  Uric Acid - High: number analyzed (Participants) | 6 | 8 | 7 | 8
  Uric Acid - High | 16.7 | 12.5 | 0 | 0
  Creatinine Clearance - Low: number analyzed (Participants) | 6 | 7 | 8 | 7
  Creatinine Clearance - Low | 16.7 | 0 | 0 | 0
  Creatinine Clearance - High: number analyzed (Participants) | 3 | 3 | 5 | 3
  Creatinine Clearance - High | 66.7 | 33.3 | 20.0 | 33.3

25. Primary Outcome: Part 2: Percentage of Chronic Hepatitis B Participants With Laboratory Abnormalities Based on Hematology, Clinical Chemistry, Coagulation and Urinalysis Test Results
Description: as for outcome 23
Time Frame: From randomization up to Week 12
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohorts 1-3: Placebo | Part 2: Cohort 1 and 2 | Part 2: Cohort 3 | Part 2 Cohort 4: Placebo | Part 2: Cohort 4
Number analyzed (Participants) | 6 | 16 | 8 | 5 | 15
percentage of participants
  Eosinophil Absolute - High: number analyzed (Participants) | 6 | 16 | 8 | 0 | 0
  Eosinophil Absolute - High | 0 | 6.3 | 0 |  |
  Erythrocyte Mean Corpuscular HGB Concentration - Low: number analyzed (Participants) | 0 | 0 | 0 | 5 | 15
  Erythrocyte Mean Corpuscular HGB Concentration - Low |  |  |  | 0 | 6.7
  Erythrocyte Mean Corpuscular Volume - High: number analyzed (Participants) | 6 | 15 | 6 | 0 | 0
  Erythrocyte Mean Corpuscular Volume - High | 0 | 6.7 | 0 |  |
  Hemoglobin - Low: number analyzed (Participants) | 0 | 0 | 0 | 5 | 15
  Hemoglobin - Low |  |  |  | 0 | 6.7
  Lymphocytes Absolute - Low | 16.7 | 25.0 | 25.0 | 20.0 | 13.3
  Lymphocytes Absolute - High: number analyzed (Participants) | 6 | 15 | 8 | 5 | 15
  Lymphocytes Absolute - High | 0 | 0 | 0 | 20.0 | 0
  Monocytes Absolute - Low: number analyzed (Participants) | 6 | 12 | 7 | 4 | 15
  Monocytes Absolute - Low | 16.7 | 8.3 | 14.3 | 0 | 26.7
  Monocytes Absolute - High | 16.7 | 6.3 | 0 | 0 | 0
  Neutrophils, Total, Absolute - Low: number analyzed (Participants) | 5 | 14 | 8 | 5 | 13
  Neutrophils, Total, Absolute - Low | 20.0 | 35.7 | 62.5 | 0 | 46.2
  Neutrophils, Total, Absolute - High | 0 | 6.3 | 0 | 0 | 0
  Platelet - Low | 0 | 18.8 | 12.5 | 0 | 6.7
  Red Blood Cell Count - Low | 0 | 0 | 12.5 | 0 | 6.7
  Reticulocytes, Pct - High: number analyzed (Participants) | 6 | 16 | 8 | 0 | 0
  Reticulocytes, Pct - High | 0 | 6.3 | 12.5 |  |
  White Blood Cell Count - Low: number analyzed (Participants) | 5 | 13 | 7 | 5 | 14
  White Blood Cell Count - Low | 20.0 | 46.2 | 42.9 | 20.0 | 50.0
  White Blood Cell Count - High | 0 | 6.3 | 0 | 0 | 0
  Bicarbonate CO2 - Low: number analyzed (Participants) | 5 | 16 | 8 | 5 | 14
  Bicarbonate CO2 - Low | 0 | 6.3 | 12.5 | 20.0 | 7.1
  Bicarbonate CO2 - High | 0 | 6.3 | 0 | 0 | 6.7
  Bilirubin - High: number analyzed (Participants) | 6 | 16 | 8 | 5 | 14
  Bilirubin - High | 0 | 6.3 | 0 | 0 | 7.1
  Blood Glucose, Fasting - Low | 16.7 | 12.5 | 0 | 20.0 | 0
  Blood Glucose, Fasting - High: number analyzed (Participants) | 6 | 14 | 8 | 5 | 14
  Blood Glucose, Fasting - High | 16.7 | 35.7 | 0 | 0 | 14.3
  Blood Urea Nitrogen - High: number analyzed (Participants) | 6 | 15 | 8 | 5 | 15
  Blood Urea Nitrogen - High | 33.3 | 26.7 | 12.5 | 0 | 6.7
  Calcium - Low | 0 | 6.3 | 0 | 0 | 6.7
  Chloride - Low: number analyzed (Participants) | 6 | 15 | 8 | 5 | 15
  Chloride - Low | 0 | 13.3 | 0 | 0 | 0
  Chloride - High | 16.7 | 0 | 0 | 20.0 | 0
  Cholesterol - High: number analyzed (Participants) | 3 | 14 | 8 | 5 | 8
  Cholesterol - High | 0 | 14.3 | 25.0 | 80.0 | 12.5
  Creatinine - High: number analyzed (Participants) | 5 | 14 | 8 | 5 | 15
  Creatinine - High | 0 | 7.1 | 0 | 20.0 | 0
  Cystatin C - High: number analyzed (Participants) | 5 | 15 | 8 | 5 | 15
  Cystatin C - High | 20.0 | 26.7 | 0 | 0 | 6.7
  Indirect Bilirubin - Low: number analyzed (Participants) | 6 | 16 | 8 | 4 | 15
  Indirect Bilirubin - Low | 16.7 | 18.8 | 0 | 50.0 | 53.3
  Indirect Bilirubin - High: number analyzed (Participants) | 6 | 16 | 8 | 5 | 14
  Indirect Bilirubin - High | 0 | 6.3 | 0 | 0 | 7.1
  Phosphorus - Low | 0 | 43.8 | 0 | 0 | 6.7
  Phosphorus - High: number analyzed (Participants) | 6 | 16 | 8 | 5 | 14
  Phosphorus - High | 0 | 6.3 | 0 | 20.0 | 7.1
  Potassium - High | 33.3 | 6.3 | 12.5 | 40.0 | 13.3
  Protein, Total - Low | 0 | 0 | 0 | 0 | 6.7
  Protein, Total - High: number analyzed (Participants) | 6 | 15 | 8 | 5 | 15
  Protein, Total - High | 0 | 6.7 | 12.5 | 20.0 | 0
  SGOT/AST - High: number analyzed (Participants) | 5 | 15 | 8 | 5 | 14
  SGOT/AST - High | 0 | 6.7 | 0 | 0 | 42.9
  SGPT/ALT - High: number analyzed (Participants) | 6 | 16 | 8 | 4 | 11
  SGPT/ALT - High | 16.7 | 6.3 | 0 | 25.0 | 36.4
  Sodium - High | 0 | 0 | 12.5 | 20.0 | 0
  Triglycerides, Fasting - High: number analyzed (Participants) | 6 | 14 | 8 | 4 | 14
  Triglycerides, Fasting - High | 16.7 | 50.0 | 12.5 | 50.0 | 14.3
  Uric Acid - High: number analyzed (Participants) | 6 | 15 | 8 | 5 | 14
  Uric Acid - High | 0 | 6.7 | 12.5 | 0 | 14.3
  Activated Partial Thromboplastin Time - High: number analyzed (Participants) | 6 | 15 | 7 | 4 | 15
  Activated Partial Thromboplastin Time - High | 0 | 6.7 | 0 | 0 | 13.3
  International Normalized Ratio - High: number analyzed (Participants) | 6 | 15 | 8 | 4 | 15
  International Normalized Ratio - High | 16.7 | 0 | 0 | 0 | 14.3
  Prothrombin Time - High: number analyzed (Participants) | 5 | 13 | 7 | 3 | 12
  Prothrombin Time - High | 20.0 | 30.8 | 14.3 | 66.7 | 41.7

26. Primary Outcome: Part 1: Percentage of SAD Participants With Abnormalities in Electrocardiograph (ECG) Parameters
Description: Triplicate 12-lead ECGs were obtained after the participant has been in a supine position for at least 10 minutes. Clinically significant RO7020531-related changes included confirmation of mean QTc 500 milliseconds (msec) or 60 msec longer than the pre-dose baseline.
Time Frame: From randomization up to Day 8
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-8 SAD: Placebo | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
percentage of participants
  Average Heart Rate (12-Lead Trip.) - Low | 6.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Average Heart Rate (12-Lead Trip.) - High | 0 | 0 | 12.5 | 0 | 0 | 0 | 0 | 0 | 0
  Average PR (12-Lead Trip.) - Low: number analyzed (Participants) | 16 | 7 | 8 | 8 | 7 | 8 | 8 | 8 | 8
  Average PR (12-Lead Trip.) - Low | 0 | 0 | 0 | 12.5 | 14.3 | 0 | 0 | 0 | 0
  Average PR (12-Lead Trip.) - High: number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 6 | 8 | 8 | 8
  Average PR (12-Lead Trip.) - High | 0 | 0 | 0 | 12.5 | 0 | 0 | 0 | 12.5 | 0
  Average QRS (12-Lead Trip.) - High | 0 | 0 | 0 | 0 | 0 | 12.5 | 0 | 12.5 | 0
  Average QTcF (12-Lead Trip.) - High | 0 | 12.5 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Primary Outcome: Part 1: Percentage of MAD Participants With Abnormalities in ECG Parameters
Description: Triplicate 12-lead ECGs were obtained after the participants has been in a supine position for at least 10 minutes. Clinically significant RO7020531-related changes included confirmation of mean QTc 500 msec or 60 msec longer than the pre-dose baseline.
Time Frame: From randomization up to Day 20
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-3, MAD: Placebo | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 6 | 8 | 8 | 8
percentage of participants
  Average PR (12-Lead Trip.) - Low: number analyzed (Participants) | 6 | 7 | 8 | 8
  Average PR (12-Lead Trip.) - Low | 0 | 0 | 0 | 12.5
  Average PR (12-Lead Trip.) - High: number analyzed (Participants) | 5 | 7 | 7 | 8
  Average PR (12-Lead Trip.) - High | 0 | 14.3 | 14.3 | 0

28. Primary Outcome: Part 2: Percentage of Chronic Hepatitis B Participants With Abnormalities in ECG Parameters
Description: Triplicate 12-lead ECGs were obtained after the participant has been in a supine position for at least 10 minutes. Clinically significant RO7020531-related changes included confirmation of mean QTc 500 msec or 60 msec longer than the pre-dose baseline.
Time Frame: From randomization up to Week 12
Population: Safety analysis population included all participants who had received at least 1 dose of study drug. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohorts 1-3: Placebo | Part 2: Cohort 1 and 2 | Part 2: Cohort 3 | Part 2 Cohort 4: Placebo | Part 2: Cohort 4
Number analyzed (Participants) | 6 | 16 | 8 | 5 | 15
percentage of participants
  Average Heart Rate (12-Lead Trip.) - High | 0 | 0 | 0 | 0 | 6.7
  Average PR (12-Lead Trip.) - Low: number analyzed (Participants) | 6 | 16 | 8 | 4 | 15
  Average PR (12-Lead Trip.) - Low | 0 | 0 | 0 | 0 | 6.7
  Average PR (12-Lead Trip.) - High: number analyzed (Participants) | 5 | 16 | 6 | 5 | 14
  Average PR (12-Lead Trip.) - High | 0 | 0 | 0 | 20.0 | 0
  Average QTcF (12-Lead Trip.) - Low | 0 | 6.3 | 0 | 0 | 0
  Average QTcF (12-Lead Trip.) - High: number analyzed (Participants) | 6 | 16 | 8 | 5 | 14
  Average QTcF (12-Lead Trip.) - High | 16.7 | 0 | 0 | 0 | 7.1

29. Primary Outcome: Part 1: Percentage of SAD Participants With Abnormalities in Vital Signs
Description: Vital signs include blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure, respiratory rate and pulse rate were obtained after the participant had been in a supine or sitting position for at least 5 minutes. Blood pressure measurement were performed in triplicate (can be as short as 20 second to 1 minute interval between measurements).
Time Frame: From randomization up to Day 8
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-8 SAD: Placebo | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
percentage of participants
  Average Diastolic BP - High | 0 | 12.5 | 25.0 | 0 | 0 | 0 | 0 | 0 | 0
  Average Systolic BP - High | 6.3 | 0 | 0 | 12.5 | 12.5 | 12.5 | 0 | 0 | 0
  Pulse Rate - Low | 6.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse Rate - High | 0 | 0 | 12.5 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory Rate - High: number analyzed (Participants) | 15 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 8
  Respiratory Rate - High | 26.7 | 0 | 28.6 | 0 | 0 | 0 | 12.5 | 25.0 | 0
  Temperature - Low: number analyzed (Participants) | 7 | 1 | 4 | 0 | 2 | 2 | 5 | 5 | 5
  Temperature - Low | 71.4 | 100.0 | 100.0 |  | 100.0 | 100.0 | 100.0 | 80.0 | 40.0
  Temperature - High | 12.5 | 0 | 12.5 | 0 | 0 | 0 | 0 | 25.0 | 0

30. Primary Outcome: Part 1: Percentage of MAD Participants With Abnormalities in Vital Signs
Description: as for outcome 29
Time Frame: From randomization up to Day 20
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-3, MAD: Placebo | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3
Number analyzed (Participants) | 6 | 8 | 8 | 8
percentage of participants
  Average Diastolic BP - High | 0 | 0 | 0 | 12.5
  Average Systolic BP - High | 0 | 25.0 | 12.5 | 12.5
  Pulse Rate - High | 0 | 0 | 0 | 12.5
  Respiratory Rate - High | 33.3 | 25.0 | 37.5 | 50.0
  Temperature - Low: number analyzed (Participants) | 3 | 4 | 4 | 4
  Temperature - Low | 100.0 | 100.0 | 75.0 | 50.0
  Temperature - High | 0 | 0 | 25.0 | 37.5

31. Primary Outcome: Part 2: Percentage of Chronic Hepatitis B Participants With Abnormalities in Vital Signs
Description: as for outcome 29
Time Frame: From randomization up to Week 12
Population: as for outcome 28
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohorts 1-3: Placebo | Part 2: Cohort 1 and 2 | Part 2: Cohort 3 | Part 2 Cohort 4: Placebo | Part 2: Cohort 4
Number analyzed (Participants) | 6 | 16 | 8 | 5 | 15
percentage of participants
  Average Diastolic BP - High: number analyzed (Participants) | 6 | 14 | 8 | 5 | 15
  Average Diastolic BP - High | 33.3 | 35.7 | 12.5 | 60.0 | 6.7
  Average Systolic BP - High | 50.0 | 31.3 | 12.5 | 20.0 | 6.7
  Pulse Rate - Low | 0 | 0 | 0 | 0 | 6.7
  Pulse Rate - High | 0 | 0 | 0 | 40.0 | 40.0
  Respiratory Rate - High | 16.7 | 6.3 | 12.5 | 0 | 6.7
  Temperature - Low: number analyzed (Participants) | 0 | 6 | 1 | 4 | 7
  Temperature - Low |  | 100.0 | 100.0 | 100.0 | 100.0
  Temperature - High | 0 | 12.5 | 0 | 0 | 20.0

ADVERSE EVENTS:
Time Frame: From Randomization to End of Study (up to 4.5 years)
Description: Safety analysis population included all HVs or participants who had received at least 1 dose of the study drug.
Arm/Group | Part 1 Cohorts 1-8 SAD: Placebo | Part 1 SAD: Cohort 1 | Part 1 SAD: Cohort 2 | Part 1 SAD: Cohort 3 | Part 1 SAD: Cohort 4 | Part 1 SAD: Cohort 5 | Part 1 SAD: Cohort 6 | Part 1 SAD: Cohort 7 | Part 1 SAD: Cohort 8 | Part 1 Cohorts 1-3, MAD: Placebo | Part 1 MAD: Cohort 1 | Part 1 MAD: Cohort 2 | Part 1 MAD: Cohort 3 | Part 2 Cohorts 1-3: Placebo | Part 2: Cohort 1 and 2 | Part 2: Cohort 3 | Part 2 Cohort 4: Placebo | Part 2: Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/6 | 0/8 | 0/8 | 0/8 | 0/6 | 0/16 | 0/8 | 0/5 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/6 | 0/8 | 0/8 | 0/8 | 0/6 | 0/16 | 0/8 | 0/5 | 1/15
Other Adverse Events (participants affected / at risk) | 5/16 | 2/8 | 4/8 | 2/8 | 2/8 | 2/8 | 2/8 | 2/8 | 3/8 | 5/6 | 6/8 | 7/8 | 7/8 | 3/6 | 11/16 | 6/8 | 3/5 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohorts 1-8 SAD: Placebo (N=16) | Part 1 SAD: Cohort 1 (N=8) | Part 1 SAD: Cohort 2 (N=8) | Part 1 SAD: Cohort 3 (N=8) | Part 1 SAD: Cohort 4 (N=8) | Part 1 SAD: Cohort 5 (N=8) | Part 1 SAD: Cohort 6 (N=8) | Part 1 SAD: Cohort 7 (N=8) | Part 1 SAD: Cohort 8 (N=8) | Part 1 Cohorts 1-3, MAD: Placebo (N=6) | Part 1 MAD: Cohort 1 (N=8) | Part 1 MAD: Cohort 2 (N=8) | Part 1 MAD: Cohort 3 (N=8) | Part 2 Cohorts 1-3: Placebo (N=6) | Part 2: Cohort 1 and 2 (N=16) | Part 2: Cohort 3 (N=8) | Part 2 Cohort 4: Placebo (N=5) | Part 2: Cohort 4 (N=15)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part 1 Cohorts 1-8 SAD: Placebo (N=16) | Part 1 SAD: Cohort 1 (N=8) | Part 1 SAD: Cohort 2 (N=8) | Part 1 SAD: Cohort 3 (N=8) | Part 1 SAD: Cohort 4 (N=8) | Part 1 SAD: Cohort 5 (N=8) | Part 1 SAD: Cohort 6 (N=8) | Part 1 SAD: Cohort 7 (N=8) | Part 1 SAD: Cohort 8 (N=8) | Part 1 Cohorts 1-3, MAD: Placebo (N=6) | Part 1 MAD: Cohort 1 (N=8) | Part 1 MAD: Cohort 2 (N=8) | Part 1 MAD: Cohort 3 (N=8) | Part 2 Cohorts 1-3: Placebo (N=6) | Part 2: Cohort 1 and 2 (N=16) | Part 2: Cohort 3 (N=8) | Part 2 Cohort 4: Placebo (N=5) | Part 2: Cohort 4 (N=15)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site phlebitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 4 (13)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyp (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (18) | 1 (1) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0/15 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 3 (4) | 3 (3) | 1 (1) | 3 (7) | 4 (4) | 0 (0) | 4 (4)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Premenstrual pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema ab igne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT02956850/Prot_SAP_000.pdf